CLINICAL TRIAL: NCT02564484
Title: Collection of PBMC's From Patients With Unusually Severe Vincristine-Induced Neuropathy for the Creation of Neuronal-Like Cells
Brief Title: iPSC Neurons From Adult Survivors of Childhood Cancer Who Have Persistent Vincristine-Induced Neuropathy
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Chicago (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SJLPSC; R01CA036401 (NIH)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Cancer Therapy; Pharmacogenomics; Drug Response; Genetic Variants; Vincristine-Induced Neuropathy; Cancer Survivor
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained from each cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropathy: Adult survivors who developed persistent treatment-related neuropathy.
- Control: Adult survivors who did not develop persistent treatment-related neuropathy.

SUMMARY:
This observational study is designed to establish induced pluripotent stem cells (iPSCs) from childhood cancer survivors who did or did not develop persistent treatment-induced peripheral neuropathy, from which to make human neurons for comparing their sensitivity to vincristine and other potentially neurotoxic drugs.

Investigators will assess the effects of inherited genome variations on treatment-induced peripheral neuropathy that persists in adults who were cured of childhood cancer. Cells from childhood cancer survivors who did or did not develop drug-induced neuropathy will be isolated and induced to become neurons. Cell sensitivity to anticancer agents will be tested in both groups and compared to determine if the survivors have genetic variants that correspond to those identified in companion genomic studies. This will assist in determining if gene variants increase the risk of treatment-induced neurotoxicity.

The investigators are interested in detecting changes of phenotype pre-post treatment in each group (cases, controls) respectively, as well in comparing the pre-post treatment phenotypic changes between the two groups (cases vs. controls).

DETAILED DESCRIPTION:
Participants will be recruited from an existing protocol at St. Jude (SJLIFE, NCT00760656). Complete neuropathic evaluations are obtained as part of SJLIFE, and the information will be shared for use in the SJLPSC study. A one-time blood draw will be obtained, and peripheral blood mononuclear cells (PBMC's) will be isolated for eventual creation of induced pluripotent stem cells (iPSC) that will be differentiated into human neurons. These human neurons will allow the investigators to functionally validate and further interrogate CEP72 genetic variants or variants in other genes that are associated with persistent (or acute) vincristine neuropathy using a "state of the art" cellular model of human neurons. Furthermore, creating neurons from patients at the extremes (highly sensitive to vincristine-induced neuropathy and matched controls) allows the study of differences at baseline and after treatment with vincristine.

PRIMARY OBJECTIVE:

* To establish induced pluripotent stem cells (iPSCs) from childhood cancer survivors who did or did not develop persistent treatment-induced peripheral neuropathy, from which to make human neurons to assess their sensitivity to vincristine and determine whether neurons from patients who developed neuropathy are more sensitive to vincristine or other neurotoxic chemotherapy.

SECONDARY OBJECTIVE:

* To evaluate the iPSC neurons made from patients with persistent treatment-related neuropathy and iPSC neurons from patients who did not develop neuropathy from the same treatment, for phenotypic difference prior to and after exposure to vincristine or other potentially neurotoxic medications.

ELIGIBILITY:
Inclusion Criteria - Neuropathy Patients:

* Adult survivor of childhood ALL
* Presence of any neuromotor, neurocortical, or neurocerebellar toxicity after vincristine treatment (either acute and/or persistent neuropathy)
* At least 50% of the persistent vincristine neuropathy cases will have the CEP72 promoter variant (rs924607) or a coding variant in CEP72 that is predicted to be damaging (CADD score >9). The balance of neuropathy cases will either have variants in other genes that are associated with vincristine neuropathy identified in the ongoing genome-wide association study (GWAS) of 1250 St. Jude Life ALL survivors, or have neuropathy in the absence of known genetic variants altering the risk of neuropathy.
* Patient understands the nature of the study and provides informed consent

Inclusion Criteria - Controls:

* Adult survivor of childhood diagnosis of ALL
* Absence of persistent neurotoxicity (grade 0) after completion of a standard vincristine-containing chemotherapy regimen (may or may not have experience acute neuropathy during treatment.
* Matched to a specified subject with neurotoxicity based on age (within 5 years), tumor type, chemotherapy regimen or total vincristine dosage, race and ethnicity.
* At least 50% of the controls will have the CEP72 promoter variant T/T genotype (at rs924607) or a coding variant in CEP72 that is predicted to be damaging (CADD score >9). The balance of controls will either have variants in other genes that are associated with vincristine neuropathy identified in the ongoing GWAS of 1250 St. Jude Life ALL survivors, or will not have a known genetic variant altering the risk of neuropathy.
* Patient understands the nature of the study and provides informed consent

Inclusion of Women and Minorities:

* Individuals of both genders, all races and ethnic groups are eligible for this protocol.

Exclusion Criteria - Both Cohorts:

* Treatment with other severely neurotoxic chemotherapy (i.e. cisplatin) prior to or concomitantly with vincristine. Carboplatin therapy is allowed
* Presence of peripheral neuropathy prior to vincristine therapy
* Poorly controlled or insulin-dependent diabetes or other condition likely to predispose to neurotoxicity
* Pregnant females
* Currently receiving treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases and controls for this study will be recruited from among the acute lymphocytic leukemia (ALL) survivor members of the St. Jude Lifetime Cohort study (SJLIFE). Cases will be matched for gender, tumor type, estimated cumulative vincristine dose at which toxicity occurred, intended vincristine chemotherapy regimen, age (within 5 years) and race with existing controls.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2016-02-08 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Number of participants for whom iPSCs were created | Up to 6 months after participant enrollment
  Blood will be drawn on Day 1, processed and sent to the University of Chicago for infectious diseases testing and creation of PBMCs for eventual development of iPS cells.

SECONDARY OUTCOMES:
Phenotype differences | Up to 6 months after participant enrollment
  Cell phenotypes of the iPSC neurons made from each patient (case or control) will be observed before and after treatment of neurotoxic drugs, giving for each drug a pair of observations from a patient.

CONTACTS AND LOCATIONS:
Overall Officials: William E. Evans, PharmD, Principal Investigator — St. Jude Children Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols